CLINICAL TRIAL: NCT06822257
Title: Understanding Alcohol Use in Young Adult Couples
Brief Title: Drinking in Young Adult Duos (DYAD) Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Carnegie Mellon University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Kasey Creswell, Associate Professor of Psychology; Director of Graduate Studies, Carnegie Mellon University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: AA031009; R01AA031009 (NIH)
Record Dates: First submitted 2025-01-24; First posted 2025-02-12 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Alcohol Consumption; Alcohol Drinking; Alcohol Intoxication
Keywords: alcohol administration; couples
MeSH Terms: conditions — Alcohol Drinking; Alcoholic Intoxication | interventions — Ethanol; Beverages

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Healthy couples who drink alcohol (Other): Healthy young adult couples who regularly drink alcohol
  Interventions: Drug: Alcohol beverage; Other: Non-alcohol beverage

INTERVENTIONS:
Drug: Alcohol beverage — moderate dose of alcohol
Other: Non-alcohol beverage — No alcohol given

SUMMARY:
This study examines the role of alcohol use in understanding the dynamics of romantic relationships. Couples will participate in a research session where they consume either an alcoholic or non-alcoholic beverage and complete study tasks. After the session, participants will provide information about their drinking habits, alcohol- and non-alcohol-related experiences, and relationship factors through brief surveys on their smart phones and again at 6-month and 12-month follow-up sessions. The findings from this study aim to improve understanding of alcohol use in close relationships and may inform future strategies for promoting healthier relationships and behaviors.

DETAILED DESCRIPTION:
This study investigates alcohol consumption in romantic relationships. Couples will be recruited to participate in a laboratory-based alcohol administration session, during which they will consume either a moderate dose of alcohol or a non-alcoholic beverage. Following beverage consumption, couples will complete questionnaires and tasks.

The study employs a multi-method approach to assess alcohol in couples, including self-reports and behavioral tasks, both inside and outside of the lab (e.g., using ecological momentary assessment). Additionally, participants' drinking patterns and relationship factors will be tracked over time, with follow-up assessments conducted at 6-months and 12 months post-laboratory session.

The findings from this research will provide insights into the role that alcohol consumption plays in close relationships and may inform interventions to support healthier drinking behaviors and relationship outcomes.

ELIGIBILITY:
Inclusion Criteria:

Both members of the couple must:

* be between the ages of 21 and 30
* regularly consume alcohol
* own a smartphone

Exclusion Criteria:

Neither member of the couple:

* has a history of adverse reaction to the amount of beverage used in the study
* has a history of major problems related to alcohol
* is taking medications that could adversely interact with alcohol
* is pregnant

Ages: 21 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 504 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2029-09 (Estimated); Study Completion 2029-09 (Estimated)

PRIMARY OUTCOMES:
Social behaviors-observational | During couple interactions in the lab for a total duration of 55 minutes.
  Behavioral measures of social processes using validated and reliable behavioral coding schemes to code facial expressions, speech behaviors, and speech content: the Facial Action Coding System (Ekman, Friesen, & Hagar, 2002) and the Rapid Marital Interaction Coding System (Heyman, 2004). This coding uses binary (yes/no) codes for presence/absence of behaviors at each moment in time. Higher scores represent more instances of behaviors.
Emotions | Immediately after the couple interactions in the lab referenced above.
  The 8-item Mood Measure (Fairbairn et al., 2021) will assess self-reported positive and negative emotions on scales from 0 (none) to 10 (extremely). Higher scores indicate a greater intensity of emotions.
Social behaviors-self-report | Immediately after the couple interactions in the lab referenced above.
  Participants will provide ratings of their own and their partners' social behaviors on ten-point Likert scales. Higher scores indicate a greater endorsement of each behavior.
Real-world experiences | The EMA protocol will be completed for 14 days post-lab session.
  Ecological Momentary Assessment (EMA) methods will be used to send a series of brief surveys to participants' smartphones to assess alcohol consumption (in standard alcoholic drinks).
Longer term alcohol problems | Assessed longitudinally up to 12-months post-lab session.
  Follow-up sessions will assess alcohol problems using DSM-5 alcohol use disorder criteria. Higher scores reflect more alcohol problems.

SECONDARY OUTCOMES:
Relationship functioning | Assessed longitudinally up to 12-months post-lab session.
  Relationship functioning will be assessed on 10 point Likert scales (Jakubiak & Feeney, 2009), with higher scores representing higher relationship functioning.

CONTACTS AND LOCATIONS:
Locations (1):
- Carnegie Mellon University, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared in the NIAAA Data Archive